CLINICAL TRIAL: NCT02416817
Title: Clinical Trial: Evaluation of 2 Different Protocols of Blood Derivates Transfusion in Acute Trauma Patients in a Brazilian Tertiary Hospital
Brief Title: Strategy of Transfusion in Trauma Patients - STATA Trial
Acronym: STATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STATA
Record Dates: First submitted 2014-08-28; First posted 2015-04-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2015-11

CONDITIONS: Wounds and Injuries
Keywords: Thrombelastography; Massive Transfusion; Major Trauma; Blood products; Thromboelastometry
MeSH Terms: conditions — Wounds and Injuries | interventions — Erythrocyte Count; Platelet Count; prothrombin complex concentrates; Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood Products only. (Experimental): This arm will receive 1:1:1 Red blood cells : Fresh Frozen Plasma : Platelets upon a major trauma triggers. 1:1:1 Ratio for packs of blood products. The patient will be re-evaluated every hour again for the major bleeding triggers and another 1:1:1 intervention may or may not occur.
  Interventions: Other: Blood Products only
- Point of care guided (Experimental): This arm will receive Red blood cells, Human Fibrinogen and Prothrombinic complex concentrates (PCC) based on thromboelastometry. The dosis of each drug will be determined by the analyses of the thromboelastometry curves.
  Interventions: Other: Point of Care guided

INTERVENTIONS:
Other: Blood Products only — Based solely on massive transfusion triggers Patients with traumatic hemorrhage that fulfil the inclusion criteria will receive blood products by prescription of the patient's anesthesiologist. The patient will be constantly observed and bleeding triggers will be reassessed hourly.
  Other Names: Red blood cells; Platelets; Fresh frozen plasma
  Arms: Blood Products only.
Other: Point of Care guided — Based on massive transfusion triggers and thromboelastometry Patients with traumatic hemorrhage that fulfil the inclusion criteria will receive the drugs guided by the results of the thromboelastometry. The dosis of each drug will be based on the analysis of the thromboelastometry curves (established algorithm).
  Other Names: Red blood cells; Beriplex® P/N (CSL Behring GmbH, Marburg, Germany); Haemocomplettan® P (CSL Behring, Marburg, Germany); Prothrombin Complex Concentrates (PCC); Human Fibrinogen
  Arms: Point of care guided

SUMMARY:
The purpose of this study is to compare two already validated methods for massive transfusion in trauma patients admitted to the emergency room of a large reference hospital.

DETAILED DESCRIPTION:
In this randomized trial trauma patients in need of massive transfusion will be assigned to one of the following transfusion strategies:

1. - Fresh Frozen Plasma, Platelets Concentrate and Packed red blood cells in 1:1:1 ratio.
2. - These patients will receive Red blood cells based on Haemoglobin measurements and will receive either Beriplex® P/N (CSL Behring GmbH, Marburg, Germany) or Haemocomplettan® P (CSL Behring, Marburg, Germany), or Platelets based on thromboelastometry.

To be included patients must meet the following inclusion criteria:

1. - Trauma victims
2. - Adults between 18 - 80 years old
3. - Injury Severity Score (ISS) between 15 and 45
4. - Assessment of Blood Consumption (ABC) Score ≥ 3 points
5. - Shock Index ≥ 1,2
6. - Acute hemorrhage of more than 50% estimated blood volume in 3 hours or more than 1,5 ml/kg/min of blood during 20 minutes.

Exclusion Criteria:

1. - Early cardiac arrest
2. - Pregnancy
3. - Injury Severity Score (ISS) > 45
4. - Patient transferred from another hospital
5. - Drug abuse history
6. - Known coagulation impairment
7. - Known use of anticoagulants, or platelet antiaggregants.

The group of health-care providers recruiting the patients based on eligibility criteria, is different than the group that evaluates the clinical outcomes of the included patients, in such a way that no researcher is tasked with post-randomisation care of the subjects. This is done to prevent observational bias.

Two informed consent forms are signed for each patient. The first one is signed by an independent physician. Another consent form is signed by the patient's family or the own patient within 24 hours of hospital admission.

The randomisation is performed by sealed envelopes assigned to the eligible patients anytime they reach the protocol criteria. The envelopes were created using a computer generated randomisation table specifically designed to this study.

An interim analysis was performed in October 2015 and it showed that there was no increased mortality or morbidity within the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Trauma victims
* Adults between 18 - 80 years old
* Injury Severity Score (ISS) between 15 and 45
* Assessment of Blood Consumption (ABC) Score ≥ 3 points
* Shock Index ≥ 1,2

Exclusion Criteria:

* Early cardiac arrest
* Pregnancy
* ISS > 45
* Patient transferred from another hospital
* Drug abuse history
* Known coagulation impairment
* Known use of anticoagulants, or platelet anti-aggregants. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
SOFA Score - 5 days | 5 days
  Evaluation of the SOFA score along the first 5 days after the patient admission.

CONTACTS AND LOCATIONS:
Overall Officials: Roseny R Rodrigues, M.D., Study Director — Hospital das Clínicas HC-FMUSP
Locations (1):
- Hospital das Clínicas FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data collected can be shared if needed.

REFERENCES:
- [Derived] Brunskill SJ, Disegna A, Wong H, Fabes J, Desborough MJ, Doree C, Davenport R, Curry N, Stanworth SJ. Blood transfusion strategies for major bleeding in trauma. Cochrane Database Syst Rev. 2025 Apr 24;4(4):CD012635. doi: 10.1002/14651858.CD012635.pub2. PMID 40271704